CLINICAL TRIAL: NCT05279053
Title: Mapping Brain Glutamate in Humans: Sex Differences in Cigarette Smokers
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Edythe London, Professor In Residence, University of California, Los Angeles
Other Study IDs: 17-000387
Record Dates: First submitted 2022-02-23; First posted 2022-03-15 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Cigarette Smoking; Tobacco Dependence; Sex
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use Disorder; Coitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male
- Female

SUMMARY:
The proposed study will evaluate sex differences in whole-brain glutamate (Glu), with a focus on the dorsal anterior cingulate cortex (dACC), anterior insula, and thalamus, as well as how it is influenced by sex (males vs. females), smoking state (overnight abstinent vs. sated), and circulating ovarian hormones (estrogen and progesterone) in women. Glu will be measured in almost the entire brain, with special focus on the dorsal anterior cingulate cortex (dACC), anterior insula, and thalamus, all of which have been implicated in behavioral states linked to tobacco withdrawal, using an echo-planar spectroscopic imaging (EPSI) variant of magnetic resonance spectroscopy (MRS). Serum ovarian hormones (estrogen and progesterone) will be measured for female participants to determine relationships between brain Glu and this hormone. Whole-brain Glu will be measured in 60 smokers (30 men, 30 women) twice, after overnight (~12 h) abstinence and after participants smoke the first cigarette of the day.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identified as only male or female
2. Age 18-45 years (children <18 years will be excluded due to low prevalence of conventional cigarette smoking; female participants >45 years of age will be excluded to avoid effects of perimenopause and menopause in women; male participants >45 years of age will be excluded as well to ensure that male and female groups are matched on age
3. English fluency demonstrated by verbal skills sufficient to participate in a conversation, including the ability to ask and answer questions at a level that assures adequate understanding of the study (a comprehension quiz will be given)
4. Right handedness (evaluated using the Edinburgh Inventory)
5. Generally in good health without cardiovascular, hepatic, renal, or autoimmune diseases, diabetes, or cancer
6. Must have smoked for ≥1 year
7. Must endorse inhaling while smoking
8. Must smoke ≥10 cigarettes per day
9. Must have expired CO >10 ppm and urinary cotinine ≥100 ng/ml at screening/intake
10. Fulfillment of DSM-5 criteria for Tobacco Use Disorder

Exclusion Criteria:

1. Seeking treatment for nicotine dependence within 3 months of screening
2. Medical condition that may compromise safety (based on history, physical exam)
3. Neurological disorder that would compromise compliance and/or informed consent
4. Major psychiatric disorder (e.g., Major Depression, Schizophrenia, Bipolar Disorder) per DSM-5 MINI
5. Current drug use disorders other than Tobacco Use Disorder (as defined in DSM-5)
6. Recent use of cocaine, opiates, benzodiazepines, or amphetamines as shown by urine test at the screening or testing sessions
7. Smoke marijuana >3X/week (self-report) or positive marijuana urine test on a scan day (positive at screening allowed)
8. Use of tobacco in forms other than cigarettes (e.g., snuff, chewing tobacco, e-cigarettes) >10 days in the month before screening
9. Preference for menthol cigarettes, given sex differences in the effect of menthol on the rate of nicotine entry into the brain
10. Pregnancy or nursing
11. Presence in the body of metal that would compromise safety during MRI
12. Claustrophobia
13. Any other condition that would compromise safety

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Sixty adult daily smokers (30 men and 30 women; 18-45 years old), who are otherwise in good health. Interested individuals will be invited to participate in the research project regardless of sex, race or ethnicity, although strong efforts will be made to recruit equal numbers of male and female participants. Individuals will not be excluded from study participation based on race/ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Circulating Ovarian Hormone: Estrogen - in overnight abstinent smokers | Measured before and after smoking a cigarette across a period of 2 hours
  Estrogen assayed via a blood sample
Circulating Ovarian Hormone: Progesterone - in overnight abstinent smokers | Measured before and after smoking a cigarette across a period of 2 hours
  Estrogen assayed via a blood sample
Whole Brain Glutamate | Measured before and after smoking a cigarette across a period of 2 hours
  Measured by EPSI acquisition in overnight abstinent smokers
Nicotine Metabolite Ratio | Measured before smoking a cigarette at a single timepoint
  Measured by blood sample

SECONDARY OUTCOMES:
Urge to Smoke Scale (UTS) | Measured before and after smoking a cigarette across a period of 2 hours
  This is a 10-item self-reporting questionnaire that measures cigarette craving
Shiffman-Jarvik Withdrawal Scale (SJWS) | Measured before and after smoking a cigarette across a period of 2 hours
  This is a 25-item self-reporting questionnaire that measures psychological withdrawal
Positive and Negative Affect Schedule (PANAS) | Measured before and after smoking a cigarette across a period of 2 hours
  This is a 20-item self-reporting questionnaire that measures positive and negative affect
Spielberger State-Trait Anxiety (STAI) | Measured before and after smoking a cigarette across a period of 2 hours
  This is a 20-item self-reporting questionnaire that measures anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Edythe London, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States